CLINICAL TRIAL: NCT00196690
Title: Treatment With Donepezil of Chronic Aphasia and Sensorimotor Deficits Associated to Cerebrovascular Accidents: a Double-Blind,Placebo-Controlled, Randomized Parallel Trial.
Brief Title: Donepezil in Chronic Poststroke Aphasia: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gabinete Berthier y Martínez (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-0509
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Stroke; Aphasia
Keywords: Aphasia; Donepezil
MeSH Terms: conditions — Stroke; Aphasia | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
* Aphasia (impairment of language function due to brain damage)may be treated with speech-language therapy and drugs. Several drugs have been studied but with limited success.
* Recent data suggest that the neurotransmitter acetylcholine may be reduced in brain damaged subjects and that drugs that stimulates acetylcholine activity may help recovery of aphasic deficits particularly when paired with speech-language therapy.
* Recent evidence indicates that medicaments acting on the neurotransmitter acetylcholine may promote improvement of aphasic deficits and our previous open-label study of donepezil in post-stroke aphasia showed benefits in all patients and observed benefit were long-lasting (6 months).This study will test the safety and efficacy of donepezil (an agent acting on acetylcholine)in subjects with stroke-related chronic aphasia (more than 1 yr of evolution).

DETAILED DESCRIPTION:
* Prior clinical information of donepezil treatment of post-stroke aphasia comes from single-case studies, small case-series and an open-label study. In addition, an extension phase of a small open-label study also suggest that the efficacy of donepezil in chronic post-stroke apahsia is maintained at long-term follow-up. These data collectively suggest that in post-stroke donepezil is effective and well-tolerated with a limited potential for causing clinically significant interactions when prescribed with other medications. However, these results are preliminary and should be judged parsimoniously until randomized controlled trials will be performed.Moreover, recent data by our group also showed that donepezil may improve sensorimotor deficits (hemiparesis)in some patients.
* The use of acetylcholinesterase inhibitors such as donepezil in post-stroke may be justified because in vivo and postmortem studies have shown that patients with vascular dementia and lesions in subcortical and cortical structures have deficient cholinergic neurotransmission that results from interruption of cholinergic pathways linking the basal forebrain with the cerebral cortex, including the perisylvian language area.In addition, two large-scale randomized controlled trials in patients pure vascular dementia and vascular cognitive impairment found that donepezil was significantly superior to placebo on cognition, global function and activities of daily living.And the most noticeable benefits of donepezil over placebo at doses of 5-mg and 10-mg were found on the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog/11), an assessment instrument highly reliant upon language variables (6 out of 11 items).
* We evaluated the efficacy of donepezil in patients with chronic aphasia associated with stroke.This is a 20-week, randomized, placebo-controlled, double-blind parallel study that enrolled aphasic patient with more than one year of evolution. During the study all patients continued receiving two hours weekly of conventional speech-language therapy. Patients were randomized in an 1:1 ratio to donepezil, 5-mg/day, for the first 4 weeks, followed by forced dose escalation to 10-mg/day thereafter (n =13), or placebo (n = 13) and then a 4 week washout period. The primary efficacy measures were the Aphasia Quotient (AQ) of the Western Aphasia Battery and the Communicative Activity Log. Secondary efficacy measures included selected subtests of the Psycholinguistic Assessment of Language Processing in Aphasia that examined phonological and lexical-semantic domains and the Stroke Aphasia Depression Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Chronic aphasia of more than one year duration. Must be able to complete protocol.

Exclusion Criteria:

* Heart block
* Bronchial Asthma
* Hypersensitivity to donepezil
* Dementia
* Major psychiatric illness

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Language function (overall aphasia severity)
Communication

SECONDARY OUTCOMES:
Depression
Cognitive evaluation of language function

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo L. Berthier, M.D., Ph.D., Principal Investigator — Gabinete Berthier y Martínez. Malaga, Spain. Centro de Investigaciones Médico-Sanitarias (CIMES), University of Malaga, Malaga, Spain
Locations (1):
- Gabinete Berthier y Martínez, Malaga, Spain. Centro de Investigaciones Médico-Sanitarias (CIMES), UNiversity of Malaga, Malaga, Spain., Málaga, Malaga, Spain

REFERENCES:
- [Background] Berthier ML. Poststroke aphasia : epidemiology, pathophysiology and treatment. Drugs Aging. 2005;22(2):163-82. doi: 10.2165/00002512-200522020-00006. PMID 15733022